CLINICAL TRIAL: NCT01676857
Title: Chemokine Mechanisms in Chronic Pelvic Pain
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Praveen Thumbikat, Assistant Professor, Northwestern University
Other Study IDs: STU00030121; R01DK083609 (NIH); R01DK094898 (NIH)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Prostatitis
Keywords: chronic pain, prostatitis, pelvic pain
MeSH Terms: conditions — Prostatitis; Chronic Pain; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Expressed prostatic secretions, urine with or without cells, blood for cells and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CP/CPPS group: The Study population will include patients diagnosed with CPPS (equal numbers of CPPS IIIa and CPPS IIIb) at least 18 years of age, recruited from Northwestern urology clinical site practices. All CPPS participants will be male and will have pelvic pain symptoms. Men who are at least 18 years of age and who had been seen by a physician for symptoms of CP/CPPS within the previous 2 years will comprise the patient population
- Control group: Adult male volunteers who are male, at least 18 years of age and meet inclusion and exclusion criteria

SUMMARY:
The purpose of this study is to identify biomarkers that can be utilized in the diagnosis of chronic pelvic pain syndrome in men.

DETAILED DESCRIPTION:
Chronic pelvic pain is the hallmark of patients with chronic pelvic pain syndrome (CPPS), a non-bacterial category of prostatitis that is a significant source of morbidity in American men. The cause of CPPS is unknown and there is a lack of convenient biomarkers for diagnosis of this syndrome. This project will examine the expression of biomarkers in expressed prostatic fluid from adult men with and without a diagnosis of CPPS. Thus our specific aim is to validate the use of the chemokines MCP-1 and MIP-1alpha and mast cell tryptase as biomarkers for CPPS in humans and correlate their levels with CPPS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* CP/CPPS group inclusion criteria

Patients are eligible for the study if they meet the following criteria:

* Participant has signed and dated the appropriate Informed Consent document.
* Agreed to participate in Study procedures.
* Participant is at least 18 years of age.
* Participant reports a response of at least 1 on the pain, pressure or discomfort scale (SYM-Q, Question #1).
* Participant reports pain or discomfort in any of the 8 domains of the Male Genitourinary Pain Index (MGUPI) (items 1a, 1b, 1c, 1d, 2a, 2b, 2c, 2d).
* These CP/CPPS symptoms been present for the majority of the time during any 3 months in the previous 6 months.

Exclusion Criteria:

* Participant has an on-going symptomatic urethral stricture.
* Participant has an on-going neurological disease or disorder affecting the bladder or bowel fistula.

Participant has a history of cystitis caused by tuberculosis, radiation therapy or Cytoxan/cyclophosphamide therapy.

* Participant has augmentation cystoplasty or cystectomy.
* Participant has a history of cancer (with the exception of skin cancer).
* Participant has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc).
* Participant diagnosed with unilateral orchialgia, without pelvic symptoms.
* Participant has a history of transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation, prostate cryo-surgery, or laser procedure.

Control group exclusion criteria In addition to the exclusion criteria listed above additional criteria for control subjects are as follows.

1. In the past year, symptoms of discomfort or pain in the pelvic region for extended periods of time.
2. Volunteers who have had a urinary tract infection with a urine culture value of >100,000 CFU/ml within the past three months.
3. Volunteers treated with intravesical chemotherapy or BCG.
4. Volunteers who have had any of the following sexually transmitted diseases (STDs) - gonorrhea, chlamydia, mycoplasma or trichomonas.
5. Volunteers with inflammatory bowel disease (such as Crohn's disease or ulcerative colitis, but not irritable bowel syndrome)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Study population will include 176 adult patients diagnosed with CPPS (equal numbers of CPPS IIIa and CPPS IIIb) and 88 adult comparator controls, at least 18 years of age, recruited from Northwestern urology clinical site practices. All CPPS participants will be male and will have pelvic pain symptoms. Men who are at least 18 years of age and who had been seen by a physician for symptoms of CP/CPPS within the previous 2 years will comprise the patient population.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2010-05; Primary Completion 2018-01-31 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Correlation of cytokines/chemokines/proteins with CPPS symptoms | Over the period of a year
  Cytokines/chemokines/proteins will be correlated with symptom scores from patients in a longitudinal fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Thumbikat, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

REFERENCES:
- [Background] Desireddi NV, Campbell PL, Stern JA, Sobkoviak R, Chuai S, Shahrara S, Thumbikat P, Pope RM, Landis JR, Koch AE, Schaeffer AJ. Monocyte chemoattractant protein-1 and macrophage inflammatory protein-1alpha as possible biomarkers for the chronic pelvic pain syndrome. J Urol. 2008 May;179(5):1857-61; discussion 1861-2. doi: 10.1016/j.juro.2008.01.028. Epub 2008 Mar 18. PMID 18353390